CLINICAL TRIAL: NCT00777569
Title: Study 2: Comparisons of Nicotine-free Cigarettes, Extra Low Nicotine Cigarettes vs. Medicinal Nicotine
Brief Title: Comparisons of Nicotine-free Cigarettes, Extra Low Nicotine Cigarettes vs. Medicinal Nicotine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Dorothy Hatsukami, Ph.D. Principal Investigator, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA 013333
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2008-12

CONDITIONS: Tobacco Dependence
Keywords: Smoking; PREPS; Harm reduction; Biomarkers of tobacco exposure; Compensatory smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Harm Reduction | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extra-low nicotine cigarettes (Experimental)
  Interventions: Drug: Extra-low nicotine cigarettes
- Nicotine-free cigarettes (Experimental)
  Interventions: Drug: Nicotine free cigarettes
- Medicinal Nicotine (Active Comparator)
  Interventions: Drug: Nicotine Lozenge

INTERVENTIONS:
Drug: Nicotine free cigarettes — Quest Step 2 contains 0.05 mg nicotine
  Arms: Nicotine-free cigarettes
Drug: Extra-low nicotine cigarettes — Quest 2 cigarettes contains 0.3 mg nicotine
  Arms: Extra-low nicotine cigarettes
Drug: Nicotine Lozenge — 4 mg nicotine lozenge
  Other Names: Commit
  Arms: Medicinal Nicotine

SUMMARY:
In this study, smokers will be randomly assigned to one of three conditions for six weeks: 1) nicotine-free cigarettes (0.05mg); 2) extra low nicotine cigarettes (0.3 mg); or 3) medicinal 4 mg nicotine lozenge. The tobacco toxin profiles across these various products will be compared. The effects of these products on biomarkers of exposure and risk factors for disease, compensatory smoking, components of tobacco addiction and short-term smoking cessation will be determined. Predictors of response to these products (e.g., compensatory smoking, compliance with product use, time to lapse) will also be examined.

The following primary hypothesis will be tested: 1) Extent of tobacco toxin exposure will be greatest for the extra low nicotine cigarette and least for nicotine lozenge. Other secondary hypotheses include: 2) Compensatory smoking, as calculated by using cotinine, will be greatest for the extra low cigarette compared to the nicotine-free cigarette; 3) Greater positive subjective responses to cigarettes will be observed with extra low nicotine vs. nicotine-free cigarette; 4) Similar withdrawal symptoms and negative affect will be observed with nicotine-free cigarette and nicotine lozenge, and least withdrawal and negative affect with the extra low nicotine cigarette; 6) Least dependence and greatest motivation and self-efficacy to quit will be observed with nicotine lozenge and the greatest dependence and least motivation and self-efficacy to quit with the extra low nicotine cigarette use; 7) Shorter time to lapse will be observed with extra low nicotine vs. nicotine-free cigarettes because of extinction is likely to occur with nicotine-free cigarettes, and the longest time to lapse for nicotine lozenge because the cigarette condition groups will have experienced stronger attentional bias toward cues, and more dependence prior to the quit date and greater withdrawal after the quit date.

DETAILED DESCRIPTION:
Smokers (N=150) will be enrolled in the study and will smoke ad libitum for a period of two weeks during which time they will be assessed for baseline measurements. Subjects will then be randomly assigned to one of the three conditions (N=50). Subjects will be blinded as to whether they are assigned to the Quest nicotine-free vs. extra low nicotine condition. There are no distinguishing features between these two cigarettes. Nicotine lozenge assignment is open label. Subjects will be asked to use only their assigned study product (low nicotine, nicotine-free cigarettes or lozenge) for a period of 6 weeks. Study cigarettes will be given to them at each clinic visit and subjects will be told to smoke ad libitum. They will be provided a supply equivalent to 150% of their baseline-smoking rate to allow for compensatory smoking to occur. They will keep record of each cigarette they smoked. If they smoked cigarettes other than those assigned to them, they will be asked to notate on a sheet when that cigarette was smoked. At the end of the 6-week period, they will be asked to quit smoking and NRT.

First morning urine and fasting blood samples will be collected at baseline and 2 and 6 weeks on the study products; at 6 weeks of abstinence and the 1 month follow-up.

Counseling. In each condition, subjects will be provided brief, structured counseling that is similar in duration. The subjects in the cigarette conditions will discuss any difficulties they experienced with switching cigarettes and problem solving these obstacles. Problem solving each obstacle will be solicited from the subject. However, if no solution or limited solution is provided, the counselor will provide a standardized response for each of the obstacles confronted.

Follow-up Phase. Subjects will be followed up 1 month after the end of the 6 week abstinence period.

ELIGIBILITY:
Inclusion Criteria:

* smoking between 10-40 cigarettes daily for the past year;
* in good physical health (no unstable medical condition;
* no contraindications for medicinal nicotine;
* stable, good mental health

Exclusion Criteria:

* unwilling to use study products for 6 weeks;
* unstable medical or psychiatric condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-03; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Biomarkers for tobacco exposure measures: Carbon monoxide, cotinine, NNAL-gluc, NNN, mercapturic acids, 1-hydroxypytrene and biomarkers for cardiovascular risk: WBC, lipid profile, fibrinogen, heart rate, blood pressure. | 6 weeks
Tobacco Cessation | 12 weeks

SECONDARY OUTCOMES:
Pulmonary function | 12 weeks
Nicotine withdrawal symptoms | 12 weeks
Motivation to quit and self-efficacy | 12 weeks
Perceived risk of PREPS and cigarette evaluation | 12 weeks
Compensatory smoking | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorohty Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Univerisity of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Dermody SS, Donny EC, Hertsgaard LA, Hatsukami DK. Greater reductions in nicotine exposure while smoking very low nicotine content cigarettes predict smoking cessation. Tob Control. 2015 Nov;24(6):536-9. doi: 10.1136/tobaccocontrol-2014-051797. Epub 2014 Sep 5. PMID 25192771
- [Derived] Hatsukami DK, Kotlyar M, Hertsgaard LA, Zhang Y, Carmella SG, Jensen JA, Allen SS, Shields PG, Murphy SE, Stepanov I, Hecht SS. Reduced nicotine content cigarettes: effects on toxicant exposure, dependence and cessation. Addiction. 2010 Feb;105(2):343-55. doi: 10.1111/j.1360-0443.2009.02780.x. PMID 20078491